CLINICAL TRIAL: NCT01490151
Title: Medtronic Treat to Range (TTR) Closed-Loop Control: Tuning a Treat-to-Range Controller for the Effects of High and Low Glycemic Index Meals
Brief Title: Medtronic Treat to Range (TTR) Closed-Loop Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Bruce A. Buckingham, Director, Pediatric Endocrinology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G110143; SPO 53117 (Other Grant/Funding Number: Medtronic)
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus; Type 1 Diabetes; Metabolic and Nutritional Disorders
Keywords: Hormone; Diabetes; Mellitus; Type 1; Immune; Metabolic disorder
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Nutrition Disorders; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TTR controller (Experimental): The intervention will consist of using the TTR controller (Medtronic) for post-prandial glucose control following high and low glycemic meals
  Interventions: Device: TTR controller (Medtronic)

INTERVENTIONS:
Device: TTR controller (Medtronic) — Subjects will arrive in the morning and the TTR controller (Medtronic) will be initialized, and then they will give their usual premeal insulin bolus for breakfast. At lunch, they will either have a low glycemic index meal or a high glycemic index meal and the meal bolus will be omitted. The device will be turned off before dinner, they will have their usual insulin bolus for dinner, eat dinner, and then be discharged to home. On another admission, they will receive an insulin dose before lunch which will be 120% of their usual insulin bolus.

SUMMARY:
The purpose of this study is to evaluate a treat-to-range automated insulin management system using continuous glucose monitoring (CGM) and subcutaneous insulin pump infusion in individuals with type 1 diabetes.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the safety and efficacy of a closed-loop "treat-to-range" (TTR) system in an inpatient clinical research center setting. The TTR system only effects insulin delivery when the glucose is projected to be above or below specified target ranges. These initial studies will assess the safety of this algorithm (mathematical equation) under the extreme conditions of a missed meal insulin bolus and meal over-insulinization. This is a "hybrid" system, which allows the research team to deliver insulin boluses manually with the TTR controller only becoming active when blood glucose levels are projected to be out of the specified range.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year.
2. Age 15 years to less than 30 years old.
3. HbA1c < 10%.
4. Subject has used a downloadable insulin pump for at least 3 months.
5. Parent/guardian and subject understand the study protocol and agree to comply with it.
6. Subject comprehends written English.
7. Subject has a home computer with email access.
8. For females, subject not intending to become pregnant during the study.
9. No expectation that subject will be moving out of the area of the clinical center during the study.
10. Informed Consent Form signed by the subject or guardian.
11. Subjects cannot have had a severe hypoglycemic event described as a seizure, loss of consciousness requiring an emergency department visit or hospitalization within 6 months of enrollment.

Exclusion Criteria:

1. Asthma if treated with systemic or inhaled corticosteroids in the last 6 months; Subject has taken oral or injectable corticosteroids within the last 30 days; Current use of oral/inhaled Glucocorticoids
2. Cystic fibrosis
3. Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
4. Use of non-insulin medications that may affect blood glucose (eg Symlin),
5. Systolic blood pressure >140 on screening; Diastolic blood pressure >90 on screening
6. History of seizure or loss of consciousness in the last 6 months.
7. Adhesive allergies; Active skin condition that would affect sensor placement
8. History of heart disease
9. Active Graves disease;
10. Currently on beta blocker medication;
11. Unwilling or unable to follow the protocol;
12. History of diagnosed medical eating disorder;
13. History of known illicit drug abuse or prescription drug abuse;
14. History of current alcohol abuse;
15. History of visual impairment which would not allow subject to participate
16. Currently participating in an investigational study (drug or device);
17. Other major illness that in the judgment of the investigator might interfere with the completion of the protocol: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University and Stanford Hospital & Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TTR Controller: The intervention will consist of using the Treat to Range (TTR) controller (Medtronic) for post-prandial glucose control following high and low glycemic meals
  TTR controller (Medtronic): Subjects will arrive in the morning and the TTR controller (Medtronic) will be initialized, and then they will give their usual premeal insulin bolus for breakfast. At lunch, they will either have a low glycemic index meal or a high glycemic index meal and the meal bolus will be omitted. The device will be turned off before dinner, they will have their usual insulin bolus for dinner, eat dinner, and then be discharged to home. On another admission, they will receive an insulin dose before lunch which will be 120% of their usual insulin bolus.
Period: Overall Study
Arm/Group | TTR Controller
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects with Type 1 Diabetes
Arm/Group | TTR Controller
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety and Feasibility of TTR Closed-loop Control System as Measure by the Count of Successful Hospital Admissions
Description: A successful hospital admission was defined as requiring no more than 2 TTR closed-loop control system adjustments of algorithm tuning parameters after initial set up, and not meeting any stopping criteria. The system was considered feasible if 75% of hospital admissions were successful.
Time Frame: Day of hospital admission (12 hours)
Population: A total of 25 admissions were completed. 1 participant was admitted twice in Cohort A1, and 2 participants were admitted first in Cohort A1 and then again in Cohort B.
Measure: Count of Units; unit: Admissions
Units Other Than Participants: Admissions
Groups:
- Cohort A1 - Missed Bolus Meal: The intervention will consist of using the TTR controller (Medtronic) for post-prandial glucose control following high and low glycemic meals
  TTR controller (Medtronic): Subjects will arrive in the morning and the TTR controller (Medtronic) will be initialized, and then they will give their usual premeal insulin bolus for breakfast. At lunch, they will either have a low glycemic index meal (Cohort A1) or a high glycemic index meal (Cohort A2) and the meal bolus will be omitted. The device will be turned off before dinner, they will have their usual insulin bolus for dinner, eat dinner, and then be discharged to home. On another admission, they will receive an insulin dose before lunch which will be 120% of their usual insulin bolus (Cohort B).
- Cohort A2 - Missed Bolus Meal: The intervention will consist of using the TTR controller (Medtronic) for post-prandial glucose control following high and low glycemic meals
  TTR controller (Medtronic): Subjects will arrive in the morning and the TTR controller (Medtronic) will be initialized, and then they will give their usual premeal insulin bolus for breakfast. At lunch, they will have a high glycemic index meal and the meal bolus will be omitted. The device will be turned off before dinner, they will have their usual insulin bolus for dinner, eat dinner, and then be discharged to home.
- Cohort B - Overbolus Meal: The intervention will consist of using the TTR controller (Medtronic) for post-prandial glucose control following high and low glycemic meals
  TTR controller (Medtronic): Subjects will arrive in the morning and the TTR controller (Medtronic) will be initialized, and then they will give their usual premeal insulin bolus for breakfast. At lunch, they will receive an insulin dose which will be 120% of their usual insulin bolus. The device will be turned off before dinner, they will have their usual insulin bolus for dinner, eat dinner, and then be discharged to home.
Arm/Group | Cohort A1 - Missed Bolus Meal | Cohort A2 - Missed Bolus Meal | Cohort B - Overbolus Meal
Number analyzed (Participants) | 8 | 7 | 9
Number analyzed (Admissions) | 9 | 7 | 9
Admissions
  Successful Admission | 7 | 4 | 7
  Unsuccessful Admission | 2 | 3 | 2

ADVERSE EVENTS:
Time Frame: Day of hospital admission (12 hours)
Description: Per protocol, adverse events were only collected during the hospital admission when participants were wearing the TTR controller (Medtronic) device
Arm/Group | TTR Controller
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 6/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TTR Controller (N=22)
Significant Post-Prandial Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — Yellow Springs Instrument (YSI) Blood Glucose Value >300 mg/dL for 75 minute in 3 hours following a meal
Hypoglycemia <50 mg/dL (Metabolism and nutrition disorders) | 2 (2) — YSI blood glucose value <50 mg/dL
Hypoglycemia (Metabolism and nutrition disorders) | 6 (6) — Any hypoglycemic event requiring administration of fast acting carbohydrates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No